CLINICAL TRIAL: NCT05973500
Title: Implementing Metabolomics Informed Diet on Inflammatory Bowel Disease Patients
Brief Title: Effect of Mediterranean Diet in Inflammatory Bowel Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Monica Guma, Associate Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 800805
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mediterranean Diet (Experimental): Mediterranean Diet for 42 Days
  Interventions: Dietary Supplement: Mediterranean Diet

INTERVENTIONS:
Dietary Supplement: Mediterranean Diet — Mediterranean Diet for 42 Days

SUMMARY:
The effects of diet on inflammatory bowel disease is an under-studied area of research. The investigators are interested in further investigating the role that diet contributes to inflammatory bowel disease severity. The investigators will collect blood and stool samples from patients with inflammatory bowel disease (IBD) before and after diet changes. The stool samples will be analyzed using metabolomics and microbiome analysis to determine changes after the new diet has been implemented. The investigators will then compare changes in the patient's overall disease state by measuring markers of inflammation including C-reactive protein (CRP) and fecal calprotectin to determine how this diet affects the disease state.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Meet classification criteria for inflammatory bowel disease including those with mild to moderate Crohn's Disease as defined by a Crohn's disease activity index between 150-450, with fecal calprotectin>250, within 1 month of enrollment.

Exclusion Criteria:

* Unable to provide informed consent
* History of or current drug abuse
* Pregnancy
* Start or change in dose of standard-of-care treatment within 12 weeks of the screening
* Known allergy to any component of the proposed diet
* Subjects with significant other medical or psychiatric comorbidities and /or medication use which in
* physician's clinical judgment might difficult the interpretation of the results
* Patients that are not on a stable dose of medications, for instance, steroids, in between samples collection
* Patients on antibiotics
* Patients with C difficile infection within 4 weeks of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
short Crohn's Disease Activity Index (sCDAI) | 42 Days
  Mild to moderate Crohn's Disease is defined by a short Crohn's Disease activity index (sCDAI) between 150-450, while those in remission from Crohn's Disease have an sCDAI score below 150. An sCDAI score exceeding 450 is used as a marker of severe Crohn's Disease.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No